CLINICAL TRIAL: NCT01678300
Title: Qualitative Study of Topical Mesalamine Adherence in Patients With Ulcerative Colitis(UC)
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Alan C. Moss, Director of Translational Research, Inflammatory Bowel Disease Center, Beth Israel Deaconess Medical Center
Other Study IDs: 2012-P-000100
Record Dates: First submitted 2012-08-23; First posted 2012-09-05 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this protocol is:

1. To quantify the prevalence of adherence to topical mesalamine in patients with UC
2. To describe the determinants of medication adherence in patients with UC prescribed topical mesalamine

DETAILED DESCRIPTION:
Patient adherence with topical mesalamine is low. Behavioral and psycho-social barriers to topical mesalamine adherence exist in patients with UC. These factors can be identified using qualitative testing in order to develop and design appropriate behavioral interventions to reduce non-adherence.

The investigators will undertake an observational study of medication persistence in 100 patients in the BIDMC clinic, "Persistence Cohort". Persistence will be measured using 12-month pharmacy refill data. The investigators will also employ a qualitative research design with discrete choice modeling in two phases: Phase I - Initial Interviews with 10 patients and Phase II - Focus Groups (2) with 5 patients each.

ELIGIBILITY:
Inclusion Criteria:

* must have ulcerative colitis diagnosed by a doctor at least 1 month prior to study participation
* must be prescribed topical mesalamine (e.g. Rowasa enemas or Canasa suppositories) by a doctor
* must be receiving care at Beth Israel Deaconess Medical Center

Exclusion Criteria:

* no diagnosis of ulcerative colitis
* no prescription for topical mesalamine
* not receiving care at Beth Israel Deaconess Medical Center

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study will be adults with diagnosed Ulcerative Colitis who have been prescribed topical mesalamine (Rowasa/Canasa) for treatment of their ulcerative colitis.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of "non-persistence" amongst patients prescribed topical mesalamine for UC | 12 months

SECONDARY OUTCOMES:
Clinical outcome (remission / relapse) at 12 months grouped by persistence status | 12 months
  Clinical outcome (remission / relapse) based on Simple Colitis Activity Index Score
Adherence phenotype details | 12 months
  * Prevalence of self-reported "low adherence" amongst patients prescribed topical mesalamine
  * Demographic and disease phenotype variables associated with "non persistence" or "low adherence" using multivariate logistic regression analysis
Quality-of-life score at 12 months | 12 months
  Short Inflammatory Bowel Disease Questionnaire score at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan C Moss, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States